CLINICAL TRIAL: NCT01661296
Title: An Open Label Study of RFH Therapy as Treatment for CL Caused by Leishmania Tropica in India
Brief Title: Efficacy of Radio-frequency Induced Heat (RFH)Therapy in Treatment of Cutaneous Leishmaniasis in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sarder Patel Medical College (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Ram Awatar Bumb, Professor and Head of the Department of Dermatology, Sarder Patel Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPMC/09/10
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Cutaneous Leishmaniasis
Keywords: cutaneous leishmaniasis, heat therapy, antimony
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Hyperthermia | interventions — Diathermy; Antimony Sodium Gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium stibogluconate (Active Comparator): Intralesional SSG was administered in dose of 50 mg cm -2 of lesion once a week for 6 weeks (total six injections)
  Interventions: Drug: Sodium stibogluconate
- RFH therapy (Active Comparator): RFH therapy was administered by a single, controlled and localized delivery of radio frequencies into the lesion for 30-60 seconds under local anesthesia (1% lidocaine) using a current field radio-frequency generator (ThermoMed 1.8, Thermosurgery Inc).
  Interventions: Other: RFH therapy

INTERVENTIONS:
Other: RFH therapy — RFH therapy was administered by a single, controlled and localized delivery of radio frequencies into the lesion for 30-60 seconds under local anesthesia using a current field radio-frequency generator.
  Other Names: Heat therapy
  Arms: RFH therapy
Drug: Sodium stibogluconate — Six intralesional injections (one injection per week) of SSG 50mg/cm-2 area of lesions
  Other Names: Glucantine; SSG
  Arms: Sodium stibogluconate

SUMMARY:
Infections caused by the protozoan parasite Leishmania include cutaneous (CL), mucosal (ML) and visceral leishmaniasis (VL). Over 12 million people currently suffer from leishmaniasis, and approximately 2 million new cases occur annually, making it a major global health problem. CL CL caused by Leishmania tropica is endemic around the city of Bikaner in Thar Desert region of the State of Rajasthan . WHO recommends antimonials such as sodium stibogluconate (SSG) to treat CL. However, these drugs are toxic and have poor patient compliance as they require multiple intramuscular or intralesional injections for 3 weeks. In addition, the emergence of drug-resistant strains is rapidly increasing worldwide. We are interested in novel treatments for CL that are safe, easy to administer and effective in inducing long-term cure. Recently, radio-frequency-induced heat (RFH) therapy has been used to treat CL. This treatment involves the controlled and localized delivery of radiofrequencies into lesions for 30-60 seconds under local anesthesia. Several short-term follow-up (4-5 months) studies as well as one long-term follow-up (12 months) study involving US soldiers who were infected with L. major in Iraq found that RFH therapy was comparable, or even better, than systemic antimonials. However, more studies are needed to establish long-term efficacy of RFH therapy in treatment of CL caused by other Leishmania species that are difficult to treat with conventional drugs, and to determine the risk of disease recurrence if any in patients living in Leishmania endemic regions. The goal of this trial is to compare long term efficacy of RFH therapy in treatment of CL caused by L. tropica in patients residing in Leishmania-endemic regions of India.

DETAILED DESCRIPTION:
Study location and participants: Subjects for this study were recruited among children between the ages of 1-17 and adults between the ages of 18-85 who visit the dermatology outpatient clinic at PBM Hospital, Bikaner, with suspected CL. Informed consent was obtained from adults or from parents/legal guardians of minors for procedures and inclusion in the study. Individuals with any uncontrolled chronic medical condition, breast feeding, on immunosuppressive drugs or anticipated unavailability for follow-up were excluded from the study. Patients with more than 4 lesions were also excluded.

Study procedures: The diagnosis of CL was established by clinical examination, history of residence in an L. tropica-endemic area, and by microscopic examination of Giemsa-stained lesion smears for parasites (Leishmania tropica bodies) or lesion biopsy. For patients who were both smear and skin biopsy negative, PCR was used to detect parasites in the lesion tissue. The lesion and surrounding skin were cleaned with stabilized 0.1% chlorine dioxide solution, and local anesthesia was administered by subcutaneous injection of 2% Lidocaine around the lesion. RFH therapy was administered by a single, controlled and localized delivery of radio frequencies into the lesion for 30-60 seconds using a current field radio-frequency generator (ThermoMed 1.8; Thermosurgery Inc. USA). Patients were be prescribed an oral NSAID and topical antimicrobial cream for 5 days. Cure of infection and any recurrence was monitored by clinical follow-up at days 10 and months 1, 2, 3, 4, 6, 9, 12 and 18 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* parasitologically confirmed diagnosis of cutaneous leishmaniasis

Exclusion Criteria:

* Multiple lesions (more than 4)

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-08; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Time to heal lesion | 6 months after treatment

SECONDARY OUTCOMES:
Tissue scarring | 12 months
Recurrence/Relapse of lesion | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ram A Bumb, MD, Principal Investigator — PBM Hospital and SP Medical College, Bikaner, Rajasthan, India
Locations (1):
- PBM Hospita and SP Medical College, Bikaner, Rajasthan, India